CLINICAL TRIAL: NCT05142839
Title: Palliation of Gastric Outflow Obstruction in Case of Concomitant Biliary Obstruction. A Retrospective, Multicenter Study. (B-GOOD Study).
Brief Title: Palliation of Gastric Outflow Obstruction in Case of Concomitant Biliary Obstruction.
Acronym: B-GOOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Malignant Biliary Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-CD (Experimental): EUS-guided choledochoduodenostomy
  Interventions: Procedure: EUS-CD
- EUS-GEA (Experimental): EUS-guided gastroenterostomy
  Interventions: Procedure: EUS-GEA

INTERVENTIONS:
Procedure: EUS-CD — EUS-guided choledochoduodenostomy
  Arms: EUS-CD
Procedure: EUS-GEA — EUS-guided gastroenterostomy
  Arms: EUS-GEA

SUMMARY:
EUS-guided drainages has been largely widespread during the last 10 years, even thanks to the advent of dedicated devices, such as lumen apposing metal stents (LAMSs).

Above all, EUS-guided choledochoduodenostomy (EUS-CD) is to date considered a valuable option of treatment in case of distal malignant biliary obstruction in case of failure of endoscopic retrograde cholangiopancreatography (ERCP) due to the presence of a gastric or duodenal obstruction, unreachable papilla in case of altered anatomy, infiltrated papilla or failure of deep cannulation of the common bile duct. This modality of drainage demonstrated satisfying results, with high rate both of technical and clinical success with acceptable rate of adverse events.

When the distal malignant biliary obstruction is associated to signs and symptoms of gastric outflow obstruction (GOO) due to the presence of a gastric or duodenal stenosis, a concomitant or subsequent palliation of the stenosis may be required.

Recently, EUS-guided gastroenterostomy (EUS-GEA) has been introduced for the palliation of GOO, showing good results although technically challenging.

To date, endoscopic treatment in case of GOO, enteral stenting and EUS-GEA are possible alternatives. However, available data demonstrated that EUS-GEA seems to be superior to enteral stenting in terms of rate of reinterventions during long-term follow-up, especially when life expectancy is superior to 6 months.

However, data are lacking regarding which is the best strategy when GOO is associated to distal malignant biliary obstruction, especially when EUS-CD is performed. This is an hot topic, as it has been supposed that EUS-CD has higher rate of adverse events, especially food impaction, when a duodenal stenosis is present.

The aim of our study, therefore, is to perform a retrospective multicenter study collecting all consecutive patients affect by distal malignant biliary obstruction drained using EUS-CD, with associated GOO treated with concomitant or subsequent duodenal stenting or EUS-GEA, in order to evaluate clinical efficacy, long term outcomes and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing affected by distal malignant biliari obstruction and gastric outflow obstruction undergone EUS-CD and EUS-GEA or enteral stenting drainage between January 2016 to September 2021

Exclusion Criteria:

* Age under 18
* Enteral stenting or EUS-GEA performed before EUS-CD
* Provide an estimate of number of records you plan to review and time period that it will be covered.January 2016 to September 2021
* If the number of records you plan to exceeds 500, please provide the following:

N/A

- Provide an estimate of how long it will take you to complete the study, including the time for data analysis.

3 month for data collection and 3 weeks for data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success for EUS-CD | 6 Months
  Decreased of total bilirubin > 50% or normalization of bilirubin within 2 weeks
Clinical success for EUS-GEA and enteral stenting | 6 Months
  resolution of symptoms of GOO, with improvement in enteral diet assumption (creamy or solid) comparing to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No